CLINICAL TRIAL: NCT04898023
Title: Evaluation of Combination Zinc and Green Tea Extract Supplementation on Reduction in Symptom Duration and Severity Associated With Community Respiratory Viral Infections: a Randomized Control Trial (ZiPhenol Study)
Brief Title: Zinc and Green Tea Extract for Community Respiratory Viral Infections
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Loss of funding
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Syed Naqvi, Associate Chief Medical Officer, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2035652
Record Dates: First submitted 2021-05-18; First posted 2021-05-24 (Actual); Results first posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-02

CONDITIONS: Respiratory Viral Infection

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- zinc-green tea extract-ascorbic acid (Experimental): Randomized patients will take three (3) capsules taken orally two (2) hours following a meal twice daily x5 days and be blinded to study assignment.
  Interventions: Drug: zinc-green tea extract-ascorbic acid
- Placebo (Placebo Comparator): Randomized patients will take three (3) capsules taken orally two (2) hours following a meal twice daily x5 days and be blinded to study assignment.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: zinc-green tea extract-ascorbic acid — Compounded capsules containing each zinc citrate, green tea extract, and ascorbic acid.
  Arms: zinc-green tea extract-ascorbic acid
Drug: Placebo — Compounded capsules containing microcrystalline cellulose.
  Arms: Placebo

SUMMARY:
Zinc and green tea supplementation have both been independently studied for supporting immune health during cold and flu-like illness in non-hospitalized patients with clinical trials demonstrating promising but inconsistent results. Combination therapy may offer an improved effect as the antioxidant compounds found in green tea have been shown to increase cellular zinc concentrations thereby inhibiting viral replication. This study seeks to evaluate the effect of combination supplementation using established doses of zinc and green tea extract on symptom duration and severity from cold and flu-like illness, including COVID-19, in adult community patients enrolled in a randomized placebo-controlled trial.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, aged 18 years and older
4. Ability to take oral medication and be willing to adhere to the prescribed dosing regimen
5. Self-reported cold or flu symptoms for < 72 hours

Exclusion Criteria:

1. Pregnant or actively seeking to become pregnant
2. Positive for influenza with planned treatment with oseltamivir or baloxavir
3. Current or planned treatment with an FDA regulated drug (including those under EUA) for COVID-19
4. Chronic liver disease (i.e. baseline liver function tests (LFTs) > 1.5x the upper limit of normal (ULN) or established cirrhosis
5. Chronic renal failure stage 4 or greater
6. History of kidney stones
7. Acute secondary bacterial infection at the time of enrollment
8. Requiring hospitalization for any reason at the time of enrollment
9. History of copper or iron deficiency
10. Current prescription for quinolone antibiotics, tetracycline antibiotics, or penicillamine at the time of enrollment
11. Allergy/intolerance to any of the active ingredients under investigation including zinc citrate, green tea, and ascorbic acid (vitamin C)
12. Patients without decision making capacity
13. Currently enrolled in another clinical trial for a respiratory viral infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2022-09-21 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-12-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Missouri, Columbia, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 17 patients signed consent forms, but only 14 completed at least one study visit for which efficacy and safety endpoints could be assessed.
Period: Overall Study
Arm/Group | Zinc-green Tea Extract-ascorbic Acid | Placebo
Started | 5 | 9
Completed | 5 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zinc-green Tea Extract-ascorbic Acid | Placebo | Total
Number analyzed (Participants) | 5 | 9 | 14
Age, Continuous [Mean (Full Range); unit: years] | 19.4 [18 to 22] | 23.6 [18 to 33] | 21.5 [18 to 33]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 4 | 6 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 2 | 6 | 8
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Recovered From Cold and Flu-like Symptoms
Description: Recovery is defined as achieving a daily total symptom severity score of 0 or 1 within 7 days using an established 12 symptom scoring system, with a severity score ranging from 0-absent to 3-very severe for each symptom assessed (max of 36 points possible; higher scores indicate a greater severity of symptoms)
Time Frame: 7 days of follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Zinc-green Tea Extract-ascorbic Acid | Placebo
Number analyzed (Participants) | 5 | 9
Participants | 3 | 4

2. Secondary Outcome: Number of Patients With Self-reported Adverse Events
Description: Adverse events collected include: nausea, vomiting, indigestion, worsening of shortness of breath or difficulty breathing, allergic reaction including skin rash, and need to seek medical care (e.g. hospitalization or physician visit) for a suspected study drug related adverse effect
Time Frame: 7 days of follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Zinc-green Tea Extract-ascorbic Acid | Placebo
Number analyzed (Participants) | 5 | 9
Participants | 2 | 3

3. Secondary Outcome: Number of Patients Who Reported Days of Absence and/or Healthcare Visits
Description: Absence includes missed days from work or school and healthcare visits include hospitalization or physician office visit(s) for respiratory viral illness related complications
Time Frame: 7 days of follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Zinc-green Tea Extract-ascorbic Acid | Placebo
Number analyzed (Participants) | 5 | 9
Participants | 5 | 3

ADVERSE EVENTS:
Time Frame: 7 days for each study subject
Arm/Group | Zinc-green Tea Extract-ascorbic Acid | Placebo
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/9
Other Adverse Events (participants affected / at risk) | 2/5 | 3/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zinc-green Tea Extract-ascorbic Acid (N=5) | Placebo (N=9)
Gastrointestinal upset (Gastrointestinal disorders) | 2 (2) | 2 (2)
Allergic Reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to loss of funding this trial was stopped prior to achieving goal enrollment. As such, no conclusions can be drawn from results reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-02-23): https://cdn.clinicaltrials.gov/large-docs/23/NCT04898023/Prot_SAP_000.pdf
  • Informed Consent Form (2023-05-10): https://cdn.clinicaltrials.gov/large-docs/23/NCT04898023/ICF_001.pdf